CLINICAL TRIAL: NCT01520012
Title: Clinical Trial to Investigate the Influence of Food on Safety/Tolerability and Pharmacokinetics of YH4808 After Oral Administration in Healthy Male Subjects
Brief Title: Food Effect on Pharmacokinetics of YH4808 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH4808-102
Record Dates: First submitted 2012-01-13; First posted 2012-01-27 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
MeSH Terms: interventions — YH4808

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Sequence 1 (Experimental)
  Interventions: Drug: YH4808 100 mg
- Sequence 2 (Experimental)
  Interventions: Drug: YH4808 100 mg
- Sequence 3 (Experimental)
  Interventions: Drug: YH4808 300 mg
- Sequence 4 (Experimental)
  Interventions: Drug: YH4808 300 mg
- Sequence 5 (Experimental)
  Interventions: Drug: YH4808 300 mg

INTERVENTIONS:
Drug: YH4808 100 mg — Period1: YH4808 100 mg bid fasting condition for 7days Period2: YH4808 100 mg bid fed condition for 7days
  Arms: Sequence 1
Drug: YH4808 100 mg — Period1: YH4808 100 mg bid fed condition for 7days Period2: YH4808 100 mg bid fasting condition for 7days
  Arms: Sequence 2
Drug: YH4808 300 mg — Period1: YH4808 300 mg fasting condition Period2: YH4808 300 mg fed condition(standard meal) Period3: YH4808 300 mg fed condition(high fat meal)
  Arms: Sequence 3
Drug: YH4808 300 mg — Period1: YH4808 300 mg fed condition(high fat meal) Period2: YH4808 300 mg fasting condition Period3: YH4808 300 mg fed condition(standard meal)
  Arms: Sequence 4
Drug: YH4808 300 mg — Period1: YH4808 300 mg fed condition(standard meal) Period2: YH4808 300 mg fed condition(high fat meal) Period3: YH4808 300 mg fasting condition
  Arms: Sequence 5

SUMMARY:
The main objective is to evaluate the food effect on the pharmacokinetic profile of YH4808 100 mg b.i.d and YH4808 300 mg after oral administration in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who signed written consent after receiving thorough explanation on trial purpose, content, and characteristics of investigational drug
* Healthy male volunteers in the age between 20 to 45 years old
* Weight: over 50kg, within ±20% of ideal body weight
* Subjects who were determined to be appropriate through screening

Exclusion Criteria:

* Clinically significant disorder in liver, kidney, cardiovascular, respiratory system, endocrine system and CNS in the physical examination and clinical laboratory tests or a medical history of malignant tumor or psychological disease
* Medical history of gastrointestinal disease or acid restraining surgery, gastric/esophagus surgery (excluding appendectomy, hernia surgery)
* A history of hypersensitivity to drugs or clinically significant allergic disease
* Clinically significant abnormal values in blood chemistry(≥ 1.5 fold of normal upper limit in the levels of SGOT, SGPT)
* Subjects who had a history of drug abuse or who had a positive results on urine drug screening
* Subjects who had taken usual dose of any prescription drugs within 14 days before the treatment or who had used usual dose of OTC drugs within 7 days before the treatment(cf, be able to be enrolled in this study according to an investigatory consideration)
* Subjects who participated in another clinical trial within 2 months before enrolling in this study
* Subjects who donated whole blood within 2 months or component blood within 1 month or who are donated within 1 month before the treatment
* Subjects who drank Over 21 units/week of alcohol or subjects who were unable to stop drinking alcohol during the hospitalization
* Subjects who stopped smoking within 3 months before the treatment
* Subjects who had a beverage containing grapefruits within 24hrs before the hospitalization or who had a beverage containing grapefruits during the hospitalization
* Subjects who had a beverage containing caffeine during the hospitalization
* Subjects with clinically significant observations considered as unsuitable based on medical judgment by investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve of YH4808 | Blood sampling during 24 or 48 hrs after administration
  non-compartmental analysis
Peak plasma concentration of YH4808 | Blood sampling during 24 or 48 hrs after administration
  non-compartmental analysis

SECONDARY OUTCOMES:
Time to reach peak plasma concentration of YH4808 | Blood sampling during 24 or 48 hrs after administration
  non-compartmental analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Yuhan Corporation, Seoul, South Korea

REFERENCES:
- [Derived] Kim E, Kim A, Yi S, Kim YK, Jang SB, Byun HM, Yoon SH, Cho JY, Jang IJ, Yu KS, Lee S. Effect of food on the pharmacokinetics of YH4808, a potassium-competitive acid blocker, after single- and multiple-oral dosing in healthy subjects. Eur J Clin Pharmacol. 2018 Oct;74(10):1261-1272. doi: 10.1007/s00228-018-2502-9. Epub 2018 Jun 15. PMID 29907887